CLINICAL TRIAL: NCT00724347
Title: PC-based Rehabilitation of Auditory Function
Acronym: CINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: US Department of Veterans Affairs (U.S. Federal Agency)
Responsible Party: Sponsor
Organization: VA Office of Research and Development (U.S. Federal Agency)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: C4739-R
Record Dates: First submitted 2008-07-24; First posted 2008-07-29 (Estimated); Results first posted 2015-01-13 (Estimated); Last update posted 2015-01-27 (Estimated); Status verified 2015-01

CONDITIONS: Hearing Loss, Sensorineural
Keywords: Auditory Perception; Hearing Loss; Presbycusis; Perceptual Learning; Hearing Prosthesis; Speech Discrimination; Delayed Treatment
MeSH Terms: conditions — Hearing Loss, Sensorineural; Hearing Loss; Presbycusis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm 1 (Experimental): Hearing impaired listeners with hearing aids underwent two months of consonant identification training in their homes.
  Interventions: Behavioral: Consonant Identification Training

INTERVENTIONS:
Behavioral: Consonant Identification Training — Subjects received psychophysically adaptive, consonant identification training in consonant discrimination on PCs in their homes.

SUMMARY:
Many older subjects experience difficulty in understanding speech in noisy environments. Part of this problem is related to changes that occur in the ear with age and compromise the hearing of high-pitched sounds. Another part of the problem with speech understanding relates to changes with age in the neural circuits of the brain that process different speech sounds. Evidence suggests that these changes in neural circuits are particularly large if hearing loss is present. Thus, while hearing aids may help compensate for hearing deficits by amplifying speech sounds, additional treatment is necessary to restore optimal neural connections in the brain so that speech sounds can be accurately distinguished from each other. We are developing PC-based training programs in an attempt to restore optimal neural connections. The current randomized trial will evaluate whether two months of training to improve the ability to discriminate different consonant sounds in noise will also improve the understanding of continuous speech and enhance auditory memory and other high-level auditory functions.

DETAILED DESCRIPTION:
More than 300,000 veterans with sensorineural hearing loss (SNHL) are fitted with VA-issued hearing aids (HAs) each year with the primary goal of improving their understanding of speech. Even older veterans without hearing loss experience a gradual decline in speech discrimination due to age-related changes in auditory function that compromise speech understanding in everyday environments. Neuroplastic reorganization within the central auditory system due to SNHL and aging contribute to these effects and compromise subjects' ability to process phonetic cues that are essential for understanding speech in noise. As a consequence, even when a HA restores high frequency signals to the cochlea in a patient with SNHL, speech understanding will remain suboptimal in the absence of rehabilitative perceptual learning.

We have developed perceptual learning paradigms that drive this rehabilitative reorganization and significantly improve speech discrimination in new HA users. We now propose to test improved training paradigms in new and experienced HA users and older subjects with normal hearing. In Exp. 1 we will evaluate baseline speech discrimination in these populations using speech-reception thresholds (SRTs) in sentences, consonant-vowel-consonant nonsense syllable tests (CVC-NST), tests of tone-pattern discrimination, and tests of auditory short-term verbal memory (ASTVM). An analysis of the correlations of these measures will provide information about basic processes underlying impaired word and sentence identification. In Exp. 2 we will investigate the effects of CVC-identification training using performance-adapted masking noise. Based on our previous results, we anticipate that training will significantly improve CVC-NST scores. We will examine the extent to which training improves SRTs, tone-pattern processing, and ASTVM. In Exp. 3 we will train subjects in a tone-pattern identification task to evaluate the extent to which non-phonetic factors (e.g., familiarity with the computerized hearing tests, placebo effects of training, improvements in auditory attention, etc.) may contribute to training benefit. In Exp. 4 we will compare the benefits of training with single-consonant syllables with the benefits of two-consonant syllable training studied in Exp. 2. Finally, in Exp. 5 we will study the benefits of CVC training using consonant-specific noise levels adjusted to compensate for intrinsic differences in the discriminability of different consonants and compare them to the benefits of global adaptive training from Exp. 2. The experiments will clarify fundamental mechanisms underlying deficits in speech discrimination and ASTVM, provide insight into the nature of training-related improvements, and elucidate the parameters needed to optimize hearing rehabilitation.

Relevance to the VA patient care mission: HAs are relatively ineffective in improving the ability of hearing-impaired subjects to understand speech in many everyday listening situations. These experiments will clarify the extent to which perceptual training can improve speech discrimination and enhance ASTVM in these conditions in new and experienced HA users and older subjects with normal hearing. Perceptual training could potentially benefit millions of veterans who wear HAs as well as older veterans with normal hearing who experience difficulties in understanding and remembering speech.

ELIGIBILITY:
Inclusion Criteria:

* Older subjects with normal hearing.
* Older subjects with mild sensorineural hearing loss who have recently received hearing aids.
* Some young subjects with normal hearing for developing training paradigms.

Exclusion Criteria:

* Health problems that would preclude training.
* Dementia.

Ages: 18 Years to 78 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-07; Primary Completion 2013-03 (Actual); Study Completion 2013-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David L. Woods, PhD, Principal Investigator — VA Northern California HCS

REFERENCES:
- [Result] Woods DL, Doss Z, Herron TJ, Yund EW. Age-related changes in consonant and sentence processing. J Rehabil Res Dev. 2012;49(8):1277-91. doi: 10.1682/jrrd.2011.08.0150. PMID 23341320
- [Result] Woods DL, Yund EW, Herron TJ, Ua Cruadhlaoich MA. Consonant identification in consonant-vowel-consonant syllables in speech-spectrum noise. J Acoust Soc Am. 2010 Mar;127(3):1609-23. doi: 10.1121/1.3293005. PMID 20329860
- [Result] Woods DL, Yund EW, Herron TJ. Measuring consonant identification in nonsense syllables, words, and sentences. J Rehabil Res Dev. 2010;47(3):243-60. doi: 10.1682/jrrd.2009.04.0040. PMID 20665350
- [Result] Yund EW, Woods DL. Content and procedural learning in repeated sentence tests of speech perception. Ear Hear. 2010 Dec;31(6):769-78. doi: 10.1097/AUD.0b013e3181e68e4a. PMID 20562624

RESULTS

PARTICIPANT FLOW:
Recruitment Details: VA patients with hearing loss who wore hearing aids (HAs) were recruited from the VA audiology clinic. Control subjects of similar ages as well as young control subjects were also recruited in order to characaterize speech discrimination capabilities in normal-hearing populations.
Pre-assignment Details: Most listeners with hearing loss were tested with and without their hearing aids prior to beginning 8 weeks of at-home PC training.
Groups:
- Arm 1: PC-Based Consonant Discrimination Training: Subjects will receive adaptive training in consonant discrimination on PCs in their homes.
Period: Overall Study
Arm/Group | Arm 1
Started | 18 (Training was the final step in the program, once the outcome tests had been developed.)
Baseline Testing | 18
Completed | 16
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Hearing impaired with hearing aids
Groups:
- Training Group: Hearing impaired subjects with bilateral, symmtrical sloping hearing losses who wore hearing aids
Arm/Group | Training Group
Number analyzed (Participants) | 18
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.67 (6.51)
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 18
Region of Enrollment [Number; unit: participants]
  United States | 18
Audiometry [Mean (Standard Deviation); unit: Sound intensity dB HL] — Pure tone audiometric thresholds measured in dB HL (i.e., relative to normal hearing listeners) from 250 to 8000 Hz in each ear.
  Sound intensity dB HL
    Thresholds 500 Hz | 19.69 (13.35)
    Thresholds 1000 Hz | 29.38 (16.42)
    Thresholds 2000 Hz | 43.13 (15.15)
    Thresholds 4000 Hz | 66.88 (9.46)
    Thresholds 6000 Hz | 71.25 (12.58)

OUTCOME MEASURES:

1. Primary Outcome: .Speech Discrimination Ability
Description: Mean consonant identification threshold improvement measure in z-scores (re normal hearing subjects) on consonant and sentence discrimination tests. Additional computerized tests measured auditory short-term verbal memory, and auditory pattern discrimination. The results were compared with baseline performance in the listener group as well as performance in other older hearing impaired subjects who used hearing aids, but who did not undergo training. In the next month, we will published two manuscripts in PLoS ONE describing (1) the benefits of hearing aids on speech comprehension in the absence of perceptual training; (2) the additional benefits of perceptual training. More metholdological details can be found in those manuscripts.
Time Frame: Subjects will receive two months of PC training and be tested before and after 2-months of training with speech tests in the laboratory..
Population: older hearing impaired listeners with hearing aids.
Measure: Mean (Standard Deviation); unit: signal to noise ratio in dB SNR
Arm/Group | Training Group
Number analyzed (Participants) | 16
signal to noise ratio in dB SNR
  Improvement in consonant thresholds | 9.43 (4.84)
  Improvement in sentence thresholds | 0.46 (1.23)

ADVERSE EVENTS:
Time Frame: 4 years
Arm/Group | Arm 1
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Five publications describing the new tests that we developed have appeared.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes